CLINICAL TRIAL: NCT04520724
Title: The Production of a Functional Roll Supporting the Treatment of Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Functional Roll for Non-alcoholic Fatty Liver Disease
Acronym: NAFLDroll
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Ewa Stachowska, Professor, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WNoZ 330/04/S/17
Record Dates: First submitted 2018-07-31; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: gut microbiome; plant fiber; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): 30 patients with NAFLD which consumes rolls with a higher fiber content twice daily (ca. 300 kcal; no less than 12 g of fiber) for 8 weeks.30 patients with NAFLD which consumes rolls with a higher fiber content twice daily (12 g of fiber/per roll) for 8 weeks.
  Rolls should be eaten for 1st and 2nd breakfast. Before starting the study, patients will receive nutritional guidelines how compose a meal that the caloric content does not exceed 400 kcal per breakfast. At the beginning patients will be trained by licensed dietitians on the principles of diet in NAFLD. During 8 weeks of intervention, patients will have telephone access to consultations with a dietitian.
  Interventions: Dietary Supplement: plant fiber
- Placebo group (Placebo Comparator): 30 patients with NAFLD which consumes rolls with a lower fiber content twice daily (ca. 300 kcal; no less than 6 g of fiber) for 8 weeks.30 patients with NAFLD which consumes rolls with a lower fiber content twice daily (6 g of fiber/per roll) for 8 weeks.
  Rolls should be eaten for 1st and 2nd breakfast. Before starting the study, patients will receive nutritional guidelines how compose a meal that the caloric content does not exceed 400 kcal per breakfast. At the beginning patients will be trained by licensed dietitians on the principles of diet in NAFLD. During 8 weeks of intervention, patients will have telephone access to consultations with a dietitian.
  Interventions: Dietary Supplement: maltodextrin bar

INTERVENTIONS:
Dietary Supplement: plant fiber — The patients with NAFLD (study and control group) will receive low-processed rolls with an 12 g plant fiber content twice daily, which would be a convenient for easy replenishment of the amount of vegetable fiber (act as prebiotic) in the diet. The intervention will be preceded by a 21 day wash-out period during which subjects will be asked to avoid foods containing large amount of fiber.
  Other Names: high fiber rolls
  Arms: Study group
Dietary Supplement: maltodextrin bar — The patients with NAFLD (placebo group) will receive maltodextrin bars twice daily, which would be a convenient and easy-to-eat snack replacing the second breakfast and afternoon tea. The bars must be eaten with 180 ml of water or unsweetened liquid. The intervention will be preceded by a 21 day wash-out period during which subjects will be asked to avoid foods containing large amount of fiber.
  Arms: Placebo group

SUMMARY:
Background: Low physical activity and poor eating habits (incl. high fat and carbohydrates but low fiber intake) are the main reason of obesity epidemic in western societies. The most common clinical complication of this condition is non-alcoholic fatty liver disease (NAFLD), that can lead to liver cirrhosis and its complications. Recent studies show that gut dysbiosis may play a crucial role in the pathogenesis of NAFLD. On the other hand plant fiber shows beneficial properties in remodeling of the gut microbiome. Aim: The project aims to create low-calorie bars / snacks with an increased fiber content (12 g/bar), replacing the second breakfast and/or afternoon tea. The main scientific aim is to examine the influence of the extra supply of fiber on i. gut microbiota composition and metabolism and ii. liver function in patients with NAFLD. Methods: Randomized placebo-controlled double blind study. A group of patients diagnosed with NAFLD, divided into 2 groups: study (12% fiber bar) and placebo (maltodextrin bar). Two study phases: preliminary study (5 weeks, 20 patients) and main study (24 weeks, 120 patients). Both clinical and laboratory (stool and serum) aspects will be analyzed, incl. anthropometric measurements, nutrition tests (food frequency questionnaire), health-related quality of life, liver ultrasound and elastography, serum and stool biochemistry and microbiome analysis.

DETAILED DESCRIPTION:
Background: High percentage of the Polish suffer from overweight and obesity. According to previous report prepared for the government, the percentage of overweight and obese people in Poland was 36.6% and 16.7% respectively, which constitutes 53.3% of the adult population in Poland. This state that body mass of a statistical -adult inhabitant of Poland is over the average one, calculated for 28 countries of the European Union. It was assumed that 25% of individuals aged ≥15 years in 2015 experienced NAFLD in France, Germany, Spain and the UK.

Obesity results from unhealthy lifestyle - too high calorie intake, too little physical activity and low fiber content in the diet. The most common clinical complication of overweight and obesity is non-alcoholic fatty liver disease (NAFLD). In the United States, 20-30% of adults suffer from NAFLD, while in the European adult population the percentage varies 14-21%. In addition, 30-50% of diabetics and 93% of people with hyperlipidemia suffer from NAFLD. The incidence of NAFLD increases with age (the disease is diagnosed between 40-65 years of age predominantly), and is sex-dependent - males suffer from this disease most often compared to women. NAFLD incidence within obese patients (BMI≥30) was found to be equal to 78%. The NAFLD risk factors include: obesity, environmental factors (low physical activity, fructose in the diet) changes in the intestinal microbiome (induced by eg. too low fiber supply) epigenetic factors, insulin resistance and genetic factors So far, there is no effective drug that can be effective in NAFLD therapy. Current treatments include changes in eating habits (proper composition of meals) leading to weight loss and thus remodeling the gut microbiome, as well as adequate physical activity. One of ingredients with beneficial effects for liver structure and function (liver cells - hepatocytes) is fiber. Plant fiber is a key component of the diet, preferably regulating metabolic processes and maintaining a healthy body. This is because the plant fiber acts as a nutrient for the intestinal flora (microbiota) and it "travels" through the intestine, ensuring its good peristalsis and proper stool formation. Undigested plant fiber including xylan polysaccharides, pectin, arabinose-containing carbohydrates as vegetable pectins, cellulose, hemicellulose, resistant starch reach unchanged into the colon, where they are metabolized by intestinal microorganisms. The fiber serves as substrate for the synthesis of short-chain fatty acids (SCFAs): propionate, acetate and butyrate. Especially the latter one - butyric acid (butyrate) is considered as a potential therapeutic agent in NAFLD. Butyrate can be treated exceptionally because of its high biological activity, which includes modulations of epigenetic functions (butyrate is a histone deacetylase (HDAC) inhibitor), energy functions (70% ATP synthesis takes place in colonocytes) and functions as a G protein-coupled receptor activator (GPCR). Consequently, the content of prebiotic vegetable fiber in the diet controls the productions of butyrate. It was shown that already after 24 hours since higher fiber supply (> 30g per day), the diversity of the microbiota was higher and the SCFAs synthesis increased. Meanwhile, the amount of fiber consumed in industrialized countries is very low. It was estimated that adults in the US provide an average of 12-18 grams of dietary fiber per day. In Europe the fiber intake varies between 16-29 g/day. At the same time in African communities (Burkina Faso, Tanzania) dietary fiber intake is high providing balance within microbial milieu within the gut, thus greater SCFA synthesis and lower titre of inflammatory factors. In comparison, in Poland the average consumption of fiber in adults is 19 - 34 g / day for men and 19 - 20 g / day for women. On the other hand most of the Nutritional Societies in the world recommend fiber intake not less than 25 g / day for women and 38 g / day for men.

As a result of inappropriate diet incl. low fiber intake obese patients show disturbances in the microbiota composition and metabolism, what results in dysfunction of intestinal barrier and increases the influx of proinflammatory substances to the liver. In this way gut dysbiosis may trigger and aggravate the liver injury in NAFLD.

Aims: The project aims to create low-calorie bars / snacks with an increased fiber content (12 g / bar), which would be a convenient and easy-to-eat snack replacing the second breakfast and/or afternoon tea. The main scientific aim is to examine whether a simple correction of the diet consisting of the extra supply of fiber in NAFLD patients will improve the microbiome composition and metabolism (inc. fermentation and production of SCFA), will support the intestinal barrier and eventually improve liver function.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD diagnosis based on non-invasive assessment

Exclusion Criteria:

* other liver disease: ALD, viral hepatitis, AIH, cholestatic liver disease, Wilson's disease, hemochromatosis, hepatobiliary cancer (HCC, CCA), incl. liver cirrhosis of any aetiology
* alcohol consumption > 21 standard drinks per week in men or >14 standard drinks per week in women over at least a two-year period,
* diabetes
* pregnancy
* celiac disease
* inflammation bowel disease
* starvation, parenteral nutrition
* drugs: metformin and other antidiabetics, statins, amiodarone, methotrexate, tamoxifen, glucocorticoids, valproate, anti-retroviral agents for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
NAFLD severity assessment | 24 weeks
  Serum non-invasive NAFLD severity parameters, liver ultrasonography and elastography at enrollment and at the end-point (NAFLD. Fibrosis (scarring) and steatosis will be asses FibroScan as (FibroScan steatosis result -CAP) in decibels per meter (dB/m). Elastography (TE Transient elastography) will be asses in kPa.

SECONDARY OUTCOMES:
Gut microbiome | 24 weeks
  Changes in gut microbiota composition and metabolism (16 SrRNA bacterial genomic, bacterial metabolites) at enrollment and at the end-point ( The gut microbiota will be asses in Operational taxonomic units (OTUs). Microbiota richness and eveness will be asses in Shannon index, Chao and Simpson index.
Gut barriere permeability | 24 weeks
  Changes in gut barriere parameters permeability (SCFA, zonulin) at enrollment and at the end-point . ( gut barriere permeability will be asses in (µmol/g SCFA), and in mg/ml zonulin in stool.
Serum biochemistry | 24 weeks
  Lipid, glucose and liver biochemistry at enrollment and at the end-point (enzymes acitivity will be asses in U/l; lipids (cholesterol, LDL ch, HDL ch TG in mg/l, glucose in mg/dl). Enzymes (ALaT, ASpAT) in U/l.
Anthropometric | 24 weeks
  Changes in anthropometric (BIA, TANITA) and indirect calorimetry at enrollment and at the end-point (weight and height will be combined to report BMI in kg/m2, fatty tissue in percent).

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Stachowska, Professor, Principal Investigator — Department of Biochemistry and Human Nutrition
Locations (1):
- Pomeranian Medical University, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters HPF, Schrauwen P, Verhoef P, Byrne CD, Mela DJ, Pfeiffer AFH, Riserus U, Rosendaal FR, Schrauwen-Hinderling V. Liver fat: a relevant target for dietary intervention? Summary of a Unilever workshop. J Nutr Sci. 2017 May 8;6:e15. doi: 10.1017/jns.2017.13. eCollection 2017. PMID 28630692
- [Background] Singh S, Osna NA, Kharbanda KK. Treatment options for alcoholic and non-alcoholic fatty liver disease: A review. World J Gastroenterol. 2017 Sep 28;23(36):6549-6570. doi: 10.3748/wjg.v23.i36.6549. PMID 29085205